CLINICAL TRIAL: NCT00966654
Title: Effect of GLP - 1 (7-36 Amide) on Myocardial Function Following Coronary Artery Bypass Surgery
Brief Title: Effect of GLP - 1 (7-36 Amide) on Myocardial Function Following Coronary Artery Bypass (CABG) Surgery
Acronym: GLP-1 CABG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left JHU
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00013802
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: CABG
Keywords: CABG; Cardiac Surgical Patient
MeSH Terms: interventions — Sodium Chloride; glucagon-like peptide 1 (7-36)amide; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): Saline
  Interventions: Drug: Placebo
- GLP-1 (Active Comparator): GLP-1 (7-36) amide
  Interventions: Drug: GLP-1 (7-36) amide

INTERVENTIONS:
Drug: Placebo — 1.5 pmol/kg/min (5 ng/kg/min) saline infused continuously over 72 hours.
  Other Names: Saline
  Arms: Saline
Drug: GLP-1 (7-36) amide — 1.5 pmol/kg/min (5 ng/kg/min) GLP-1 infused continuously over 72 hours.
  Other Names: GLP-1
  Arms: GLP-1

SUMMARY:
This research is being done to see if giving a hormone called GLP-1 can improve heart function and reduce length of stay in the Cardiac Surgical Intensive Care Unit (CSICU) in people who have non-emergent coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
After CABG surgery, a condition known as hyperglycemia or high blood sugar often occurs even in patients who have never been diagnosed with diabetes. This high blood sugar can lead to complications after surgery such as infections at the site of the incision. Additionally, if there is any cardiac muscle injury either prior to or during surgery, the injured cardiac muscle can not use glucose (the body's fuel and energy source) as well as it did prior to the injury. This reduced ability to use glucose slows the cardiac muscles ability to repair itself and provide the normal pumping force and function needed to circulate the blood throughout the body. This inability to repair itself and/or provide the normal pumping force and function can make it difficult for the patient as well as increase the length of stay required in the CSICU.

GLP-1 has the ability to lower blood sugar and help cells use glucose for fuel and energy but when the blood sugar becomes low its glucose lowering ability decreases. In this study, we want to see we want to see if GLP-1 may help keep the blood sugar within normal limits and reduce or eliminate the need for insulin. We will also see whether it will help the heart recover more quickly.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age > 18 years of age
* Able to consent
* Scheduled for non-emergent coronary artery bypass graft (CABG)
* Have an ejection fraction < 35%
* Ischemic patients with Left Ventricular Dysfunction (LVD) who need a valve procedure with their CABG

Exclusion Criteria:

* Emergency coronary artery bypass graft surgery
* Patients with an ejection fraction > 35%
* Repeat or redo CABG patients
* Patients with a history of pancreatitis
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GLP-1: GLP-1 (7-36) amide
  GLP-1 (7-36) amide: 1.5 pmol/kg/min (5 ng/kg/min) saline or GLP-1 infused continuously over 72 hours.
  OR
  Placebo (saline)
Period: Overall Study
Arm/Group | GLP-1
Started | 12
Completed | 0
Not Completed | 12
Not completed — Study was terminated,PI left institution | 12

BASELINE CHARACTERISTICS:
Population: Although 12 participants were enrolled in this study, their assignment to study arm/group, if any, is unknown. The P.I. has left the institution and neither he, nor further data (if any), are available.
Groups:
- All Study Participants: GLP-1 (7-36) amide
  GLP-1 (7-36) amide: 1.5 pmol/kg/min (5 ng/kg/min) saline or GLP-1 infused continuously over 72 hours.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  Age, years (18-75) | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Systolic Function: Pulmonary Capillary Wedge Pressure
Time Frame: 2 years
Population: The raw study data is not available for this study. The study was terminated early due to the P.I.'s noncompliance with Johns Hopkins University School of Medicine Institutional Review Board Protocol and he has since left the institution. Significant efforts have been made to locate data, but it is unfortunately unavailable.
Groups:
- GLP-1: GLP-1 (7-36) amide
  GLP-1 (7-36) amide: 1.5 pmol/kg/min (5 ng/kg/min) saline or GLP-1 infused continuously over 72 hours.
- Saline: Saline
  Placebo: 1.5 pmol/kg/min (5 ng/kg/min) saline or GLP-1 infused continuously over 72 hours.
Arm/Group | GLP-1 | Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Insulin Infusion Requirements
Time Frame: 72 hours
Population: The raw study data is not available for this study. The study was terminated early due to the P.I.'s noncompliance with JHU IRB Protocol and he has since left the institution. Significant efforts have been made to locate data, but it is unfortunately unavailable.
Arm/Group | GLP-1 | Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was terminated prematurely due to the PI leaving the institution. The time frame for the Adverse Events (if collected) is unknown since no data is available.
Description: This study was terminated prematurely due to the PI leaving the institution. The data for the Adverse Events (if collected) is unknown since no data is available.
Arm/Group | GLP-1 | Saline
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes